CLINICAL TRIAL: NCT05406895
Title: Does the Use of CBCT Pre-operative Measurements Improve the Success Rate of Inferior Alveolar Nerve Block? - A Randomized Controlled Clinical Trial
Brief Title: Use of CBCT to Improve Inferior Alveolar Nerve Block Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2533
Record Dates: First submitted 2022-05-27; First posted 2022-06-07 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Inferior Alveolar Nerve; Mandibular Nerve Blocks
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: Parallel model for either CBCT guided or intra-oral technique. If the patients receive a two-stage implant placement technique then a cross-over model will be used.
Who Masked: Participant
Masking Description: The participants will be masked to which technique they are receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBCT first (Experimental): This group will receive the injection technique that is guided by pre-treatment measurements made from the 3D dental scan (CBCT) during implant placement surgery and if the implant is placed as a two-stage procedure, during the second stage implant uncovery will receive the standard injection technique. If the implant is placed as a one-stage procedure, the second visit will not apply.
  Interventions: Drug: 2% Lidocaine with 1:100,000 epinephrine
- Standard technique first (Active Comparator): This group will receive the standard injection technique first at the implant placement surgery and if the implant is placed as a two-stage procedure, during the second stage implant uncovery will receive the injection technique guided by the 3D dental scan (CBCT). If the implant is placed as a one-stage procedure, the second visit will not apply.
  Interventions: Drug: 2% Lidocaine with 1:100,000 epinephrine

INTERVENTIONS:
Drug: 2% Lidocaine with 1:100,000 epinephrine — 2% Lidocaine with 1:100,000 epinephrine will be used for administering the lower jaw anesthesia (inferior alveolar nerve block).

SUMMARY:
The study looks to compare the success rate of lower jaw anesthesia injection (inferior alveolar nerve) that is guided by pre-treatment 3D dental scan (CBCT) versus standard injection technique.

DETAILED DESCRIPTION:
A total of 200 participants will be recruited that have existing 3D dental scans (CBCT) and require an implant placement (that will be placed in a two stage procedure) in the lower jaw for which a lower jaw anesthesia injection (inferior alveolar nerve) block will be used. The participants will be randomly assigned into one of two groups. The first group will receive the injection technique that is guided by pre-treatment measurements made from the 3D dental scan (CBCT) during implant placement surgery and if implant is placed as a two-stage procedure, during the second stage implant uncovery will receive the standard injection technique. The second group will receive the standard injection technique first at the implant placement surgery and if implant is placed as a two-stage procedure, during the second stage implant uncovery will receive the injection technique guided by the 3D dental scan (CBCT). If the implant is placed as a one-stage procedure, the second visit will not apply. Following this, subjective and objective measurements on the success of the anesthesia will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients from the age 18 to 70 years old that are assigned to the 3 clinicians of the graduating class of LSUHSC School of Dentistry Post-graduate Periodontics program.
* Patients have been reported as an ASA I or ASA II patient that has never had an allergic reaction to lidocaine based on previous dental experience.
* The patient must be missing one or more mandibular teeth and is treatment planned for a mandibular implant that is placed that requires an inferior alveolar nerve block during surgery.
* Patient must have an existing CBCT scan within the last year or is planned for a CBCT scan for the purpose of dental implant treatment.

Exclusion Criteria:

* The exclusion criteria include patients that have undergone long term use or continuous use within the last week of opioids, analgesics, medications of nerve related pathology and non-steroidal anti-inflammatory drugs.
* Patients diagnosed with trismus.
* Patients that request for Nitrous and IV anesthesia
* Patients missing remaining teeth in the quadrant or having a history of endodontic treatment of the remaining teeth in the quadrant.
* Patients having endodontic or pulpal pathology in the teeth in the quadrant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Lingual nerve numbness | 3 minutes
  Numbness of tongue, numbness of lingual tissue
Lingual nerve numbness | 5 minutes
  Numbness of tongue, numbness of lingual tissue
Lingual nerve numbness | 8 minutes
  Numbness of tongue, numbness of lingual tissue
Lingual nerve numbness | 10 minutes
  Numbness of tongue, numbness of lingual tissue
Lingual nerve numbness | one hour
  Numbness of tongue, numbness of lingual tissue
Lingual nerve numbness | 2 hours
  Numbness of tongue, numbness of lingual tissue
Mental nerve numbness | 3 minutes
  Numbness of lips, numbness of buccal gingival tissue of canine
Mental nerve numbness | 5 minutes
  Numbness of lips, numbness of buccal gingival tissue of canine
Mental nerve numbness | 8 minutes
  Numbness of lips, numbness of buccal gingival tissue of canine
Mental nerve numbness | 10 minutes
  Numbness of lips, numbness of buccal gingival tissue of canine
Mental nerve numbness | 1 hour
  Numbness of lips, numbness of buccal gingival tissue of canine
Mental nerve numbness | 2 hours
  Numbness of lips, numbness of buccal gingival tissue of canine
Inferior alveolar nerve numbness | 3 minutes
  Numbness of buccal gingival tissue of molar
Inferior alveolar nerve numbness | 5 minutes
  Numbness of buccal gingival tissue of molar
Inferior alveolar nerve numbness | 8 minutes
  Numbness of buccal gingival tissue of molar
Inferior alveolar nerve numbness | 10 minutes
  Numbness of buccal gingival tissue of molar
Inferior alveolar nerve numbness | 1 hour
  Numbness of buccal gingival tissue of molar
Inferior alveolar nerve numbness | 2 hours
  Numbness of buccal gingival tissue of molar
Inferior alveolar nerve numbness | 3 minutes
  Cold endodontic test at 1st molar, 2nd molar, 1st premolar and 2nd premolar sites
Inferior alveolar nerve numbness | 5 minutes
  Cold endodontic test at 1st molar, 2nd molar, 1st premolar and 2nd premolar sites
Inferior alveolar nerve numbness | 8 minutes
  Cold endodontic test at 1st molar, 2nd molar, 1st premolar and 2nd premolar sites
Inferior alveolar nerve numbness | 10 minutes
  Cold endodontic test at 1st molar, 2nd molar, 1st premolar and 2nd premolar sites
Inferior alveolar nerve numbness | 1 hour
  Cold endodontic test at 1st molar, 2nd molar, 1st premolar and 2nd premolar sites
Inferior alveolar nerve numbness | 2 hours
  Cold endodontic test at 1st molar, 2nd molar, 1st premolar and 2nd premolar sites

SECONDARY OUTCOMES:
Pain during surgery | At the end of the procedure
  Pain during surgery will be measured using Visual Analog Scale (VAS) which is a linear scale from 0-100 with a lower number suggesting a more successful anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Louisiana State University School of Dentistry, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No